CLINICAL TRIAL: NCT04939961
Title: Effects of Hericium Erinaceus on Microbiota and Cognition in Older Adults
Brief Title: Effects of Hericium Erinaceus on Microbiota and Cognition
Acronym: HE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, assoc. prof., University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hericium erinaceus
Record Dates: First submitted 2021-06-10; First posted 2021-06-25 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Decline, Mild
MeSH Terms: conditions — Cognitive Dysfunction; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled
Who Masked: Participant, Investigator
Masking Description: Placebo and experimental capsules (A and B) were prepared by collaborator-investigator (MycoMedica). Both experimental and placebo capsules appear similar to each other in terms of colour, flavour, size, and shape to make sure that they cannot be distinguished. Information about capsules will be provided to participants and investigators at the end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hericium erinaceus (Experimental): 8 gram of mushroom Hericium erinaceus (containing 5 milligram of erinacines) per day
  Interventions: Dietary Supplement: Hericium erinaceus
- Placebo capsule (Placebo Comparator): 8 gram of allergen free corn starch per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hericium erinaceus — 6 capsules per day, 3 times two after breakfast, lunch and dinner
  Arms: Hericium erinaceus
Dietary Supplement: Placebo — 6 capsules per day, 3 times two after breakfast, lunch and dinner
  Arms: Placebo capsule

SUMMARY:
The study evaluates the effects of Hericium erinaceus on microbiota, cognition, and other health parameters in older adults. All measurements will be performed at baseline and ten weeks after daily consumptions of either Hericium erinaceus or placebo.

DETAILED DESCRIPTION:
Hericium erinaceus, a well-known edible mushroom, has numerous biological activities. Yamabushitake (Hericium erinaceus) is a mushroom that grows on both living and dead broadleaf trees. Yamabushitake is used as food in Japan and China. Hericenones and erinacines stimulate nerve growth factor synthesis, and therefore it is expected that H. erinaceus have some effects on brain functions and autonomic nervous system. Hericium was tested in several applications, such as dementia, Alzheimer's disease, Parkinson's disease, multiple sclerosis, neuropathy and neurasthenia. The ancient Chinese knew about these possibilities and used it to support mental functions and memory, concentration. It is also very good for various digestive problems, such as gastritis, stomach ulcers, heartburn, reflux and improvement of digestion.

Therefore, the aim of our study is to evaluate the effects of Hericium erinaceus on microbiota, cognition and related parameters in elderly. The stool samples will be taken at baseline and after ten weeks of daily consumption of Hericium erinaceus or placebo. In addition, cognitive tests, anthropometric measurements, and blood analysis (lipid profile, glucose levels and neurotrophic factors) will be measured at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* age 55 - 75 years

Exclusion Criteria:

* neurodegenerative disease
* organ transplantation
* allergy to fungi
* antibiotic consumption in the previous 3 months

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Assessment of the microbial community composition in feces samples using next-generation sequencing | Change from Baseline Microbiota composition at 10 weeks.
  For the assessment of the microbial community composition, DNA will be extracted from the frozen faecal samples (1-2 gram) with the commercial DNA Stool Mini Kit. A comparison of microbiota among treatments will be done with a meta-barcoding approach using ribosomal RNA markers with modified primers.

SECONDARY OUTCOMES:
cognitive function | Change from baseline Cognitive function at 10 weeks.
  Test of perception speed patterns, Test of series
brain derived neurotrophic factor | Change from baseline Brain derived neurotrophic factor levels at 10 weeks.
  serum level measured with ELISA assay
neuropeptide Y | Change from baseline Neuropeptide Y levels at 10 weeks.
  serum level measured with ELISA assay

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman M. Chemistry, Nutrition, and Health-Promoting Properties of Hericium erinaceus (Lion's Mane) Mushroom Fruiting Bodies and Mycelia and Their Bioactive Compounds. J Agric Food Chem. 2015 Aug 19;63(32):7108-23. doi: 10.1021/acs.jafc.5b02914. Epub 2015 Aug 5. PMID 26244378
- [Background] Chong PS, Fung ML, Wong KH, Lim LW. Therapeutic Potential of Hericium erinaceus for Depressive Disorder. Int J Mol Sci. 2019 Dec 25;21(1):163. doi: 10.3390/ijms21010163. PMID 31881712